CLINICAL TRIAL: NCT06916663
Title: A Prospective, Three-Arm, Assessor-Blinded Randomized Controlled Trial Comparing Upper Body Exercise, Combined Non-Weight Bearing Exercise, and Standard Care for Improving Cardiorespiratory Fitness and Supporting Wound Healing in Patients Undergoing Active Diabetic Foot Ulcer Treatment
Brief Title: RCT Comparing Upper Body vs. Combined Exercise Protocols During Active Diabetic Foot Ulcer Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al Hayah University In Cairo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DFU-EX2025-01
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Upper Body Exercise Group (UBE): (Experimental): Structured upper extremity and core exercise sessions while maintaining foot offloading.
  Interventions: Behavioral: Upper Body Exercise Protocol (UBE)
- Combined Exercise Group (CE): (Experimental): Structured non-weight bearing combined exercise including upper body, core, and modified lower extremity exercises while maintaining foot offloading.
  Interventions: Behavioral: Combined Non-Weight Bearing Exercise Protocol (CE)
- Standard Care Control Group (SC): (Active Comparator): Standard wound care without a structured exercise intervention.
  Interventions: Behavioral: Standard Diabetic Foot Ulcer Wound Care (SC)

INTERVENTIONS:
Behavioral: Upper Body Exercise Protocol (UBE) — Participants randomized to the Upper Body Exercise Group will perform a structured, supervised exercise regimen focused exclusively on the upper extremities and core muscles, while rigorously maintaining foot offloading prescribed for diabetic foot ulcers (DFU). This intervention is delivered face-to-face in hospital-based outpatient rehabilitation centers. Sessions are held three times per week for 12 consecutive weeks (total 36 sessions), with each session lasting 45-60 minutes.
  Each UBE session comprises a 10-minute warm-up on an arm ergometer at 40-50% of the participant's heart rate reserve (HRR), followed by a circuit of eight upper body and core exercises.
  Arms: Upper Body Exercise Group (UBE):
Behavioral: Combined Non-Weight Bearing Exercise Protocol (CE) — Participants in the Combined Exercise Group will engage in a structured exercise regimen that integrates upper body, core, and modified lower extremity exercises-all performed in a non-weight bearing or seated position to ensure complete offloading of the affected foot. Sessions are conducted face-to-face in hospital-based rehabilitation centers. Participants attend three sessions per week for 12 weeks (36 sessions total), each lasting 45-60 minutes.
  Each session begins with a 10-minute warm-up on an arm ergometer at 40-50% HRR.
  Arms: Combined Exercise Group (CE):
Behavioral: Standard Diabetic Foot Ulcer Wound Care (SC) — Participants assigned to the Standard Care Control Group will receive comprehensive DFU wound management in accordance with International Working Group on the Diabetic Foot (IWGDF) guidelines. This includes standard offloading strategies (using Total Contact Cast or removable cast walker), regular weekly wound assessments, and debridement if necessary. Diabetes management education is provided along with routine adjustments and monitoring of the offloading device to ensure proper healing support. No structured exercise intervention is added; however, all aspects of care such as continuous glucose monitoring and vascular assessments will be uniformly applied to allow comparison with the exercise groups.
  Arms: Standard Care Control Group (SC):

SUMMARY:
This randomized controlled trial (RCT) aims to evaluate the effectiveness of two different structured exercise interventions compared to standard care during active diabetic foot ulcer (DFU) treatment. Participants will be allocated to one of three groups: Upper Body Exercise (UBE), Combined Exercise (CE), or Standard Care Control (SC). The interventions are designed to improve cardiorespiratory fitness-as measured by changes in VO₂peak-and other secondary clinical, metabolic, vascular, inflammatory, muscular, and quality-of-life outcomes while ensuring proper offloading and wound management.

ELIGIBILITY:
Inclusion Criteria:

Age: Adults aged 18 years or older. Diagnosis: Confirmed diagnosis of Type 1 or Type 2 diabetes. Active DFU: Presence of a diabetic foot ulcer under active treatment, as documented by the wound care team.

Wound Stability: Ulcer size that meets protocol criteria (e.g., <2 cm² or ≥2 cm²) and without critical limb ischemia.

Ability to Exercise: Medical clearance from a physician to safely participate in unsupervised upper body and non-weight bearing exercises.

Compliance: Capacity and willingness to adhere to the study protocol, including scheduled exercise sessions and offloading procedures.

Glycemic Control: Stable glycemic control medications regimen for at least 4 weeks prior to enrollment.

Informed Consent: Ability to provide written informed consent.

Exclusion Criteria:

Critical DFU Complications: Ulcers with signs of critical limb ischemia, severe infection (e.g., osteomyelitis), or wound deterioration that contraindicates participation.

Cardiovascular Limitations: Unstable cardiac conditions (e.g., uncontrolled arrhythmias, recent myocardial infarction within 6 months), severe heart failure, or any other condition contraindicating exercise.

Neurological or Musculoskeletal Limitations: Conditions that significantly impair upper body or core exercise performance (e.g., severe arthritis, recent upper body injury).

Cognitive Impairment: Significant cognitive or psychiatric disorders that would limit the ability to provide informed consent or adhere to the intervention protocol.

Concurrent Participation: Enrollment in another clinical trial or exercise program that conflicts with the study protocol.

Other Medical Risks: Any other condition, as determined by the study physician, that places the participant at increased risk of adverse events during exercise (e.g., severe peripheral vascular disease not amenable to offloading).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2025-04-22 (Estimated); Primary Completion 2027-04-23 (Estimated); Study Completion 2027-04-23 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness (VO₂peak) | Baseline and at 12 weeks
  Change in VO₂peak measured using arm ergometry with validated protocols designed for patients with lower extremity limitations. VO₂peak is a key indicator of cardiovascular fitness, with improvements expected in response to the structured exercise interventions.

SECONDARY OUTCOMES:
Wound Healing - Percent Wound Area Reduction | 4, 8, and 12 weeks
  Reduction in wound area measured using digital planimetry. This quantifies improvement in wound healing by comparing wound sizes at different time point
Wound Healing - Time to Wound Closure | Recorded weekly during the 12-week intervention
  The duration in days from the start of the intervention until complete wound closure, determined through weekly assessments performed by the clinical team.
Wound Healing - Wound Recurrence Title | At 6-month follow-up
  Incidence of DFU recurrence in patients whose wounds have closed, providing an indicator of sustained wound healing.
Metabolic Control - HbA1c Levels | Baseline and 12 weeks
  Glycated hemoglobin concentration measured from blood samples to assess long-term glycemic control, which is crucial for wound healing in DFU patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Al Hayah University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No